CLINICAL TRIAL: NCT06569953
Title: Efficacy and Safety of Liposomal Bupivacaine Injection for Paravertebral Nerve Block in the Treatment of Acute and Chronic Pain After Thoracoscopic Pneumonectomy: A Multicenter, Randomized, Double-blind, Controlled Clinical Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: People's Hospital of Chongqing (Other); LanZhou University (Other); Xiangya Hospital of Central South University (Other); Shapingba District People's Hospital of Chongqing (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LBPB
Record Dates: First submitted 2024-08-13; First posted 2024-08-26 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Acute Pain; Chronic Pain; Postoperative Pain
MeSH Terms: conditions — Acute Pain; Chronic Pain; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Randomization was performed in a 1:1 ratio with the use of block randomization.SAS software (version 9.4 or higher) was used to generate the random number and the treatment group to which the random number was assigned.Assignment of Randomization Numbers Using the Interactive Web Response System (IWRS).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (liposomal bupivacaine） (Experimental): Participants randomized to the intervention arm received liposomal bupivacaine for paravertebral block before surgery.
  Interventions: Drug: Liposomal bupivacaine
- control (bupivacaine hydrochloride) (Active Comparator): Participants randomized to the intervention arm received bupivacaine hydrochloride for paravertebral block before surgery.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Liposomal bupivacaine — Participants randomized to the intervention arm received 266 mg of liposomal bupivacaine for paravertebral block before surgery.(The volume was expanded to 30 mL with normal saline).
  Arms: intervention (liposomal bupivacaine）
Drug: Bupivacaine Hydrochloride — Participants randomized to the intervention arm received 0.5% 100 mg of bupivacaine hydrochloride for paravertebral block before surgery.(The volume was expanded to 30 mL with normal saline)
  Arms: control (bupivacaine hydrochloride)

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of liposomal Bupivacaine administered by paravertebral block for the treatment of acute and chronic pain after video-assisted thoracoscopic lobectomy.

DETAILED DESCRIPTION:
Researchers will compare liposomal bupivacaine to bupivacaine to see if liposomal bupivacaine works better to treat acute and chronic pain after video-assisted thoracoscopic lobectomy.Participants will:1.Received liposomal bupivacaine or bupivacaine paravertebral block before surgery. 2.Keep a diary of their pain scores within 30min after recovery from anesthesia and 6h, 12h, 24h, 48h, 72h and 90d after the beginning of injection of experimental drugs.

ELIGIBILITY:
Inclusion Criteria:

* Participants who scheduled for elective video-assisted thoracoscopic lobectomy under general anesthesia.
* Participants were 18 years or older.
* 18 kg/m2≤BMI≤30 kg/m2
* Participants with American Society of Anesthesiology (ASA) physical status I-III.
* Understand the significance, possible benefits, potential risks of the trial in detail.Understand the procedures and methods of this study.Willing to complete the trial in strict compliance with the clinical trial protocol.Sign the informed consent form voluntarily.

Exclusion Criteria:

* with severe cardiovascular and cerebrovascular diseases such as myocardial infarction,unstable angina pectoris,severe cardiac rhythm disorders (second- and third-degree heart block,etc.), New York Heart Association (NYHA) functional class III/IV,Ischemic stroke.
* with psychiatric disorders (such as schizophrenia,depression,etc.) and cognitive impairment.
* with sensory disorders such as hyperalgesia.
* with other bodily pain.
* allergy to amide-type local anesthetics or any of the trial drugs
* taking drugs that affect liver metabolism,corticosteroids,benzodiazepines,non-steroidal anti-inflammatory drugs(NSAIDs),opioid agonist-antagonist,central-alpha 2-agonists,anticonvulsants,antidepressants within 72h.
* with a history of alcohol or opioid abuse.
* who were pregnant or lactating.
* who were currently included in another clinical study within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Area under the movement-evoked pain intensity-time curve | from 0-72 hours after the intervention
  Area under the pain intensity-time curve in the movement (or coughing) state within 72h after the intervention.
The incidence of chronic postoperative pain | postoperative day (POD) 90
  The incidence of chronic postoperative pain at 90 days

SECONDARY OUTCOMES:
Area under the rest pain intensity-time curve | from 0-72 hours after the intervention
  Area under the pain intensity-time curve at rest within 72h after the intervention.
Movement-evoked pain score | 30 minutes after recovery from anesthesia,6 hours, 12hours, 24hours , 48hours and 72 hours after the intervention
  Use pain Numeric Rating Scale(NRS) to evaluate the movement-evoked pain score at 30minutes after recovery from anesthesia and at 6 hours, 12hours, 24hours , 48hours and 72 hours after the intervention.(NRS scale 0-10, where 0 was no pain, and 10 was the worst possible pain)
Pain score at rest | 30 minutes after recovery from anesthesia,6 hours,12hours, 24hours , 48hours and 72 hours after the intervention
  Use pain Numeric Rating Scale(NRS) to evaluate the pain score at rest at 30minutes after recovery from anesthesia and at 6 hours, 12hours, 24hours , 48hours and 72 hours after the intervention.(NRS scale 0-10, where 0 was no pain, and 10 was the worst possible pain)
Proportion of participants who did not use rescue analgesia | from 0-72 hours after the intervention
  Proportion of participants who did not use rescue analgesia during 0-12 hours, 12-24 hours, 24-48 hours, 48-72 hours and 0-72 hours after the intervention.
The cumulative dosage of rescue analgesia | from 0-72 hours after the intervention
  The cumulative dosage of rescue analgesia during 0-12 hours, 12-24 hours, 24-48 hours, 48-72hours and 0-72hours after the intervention.
The time of first use of rescue analgesia | from 0-72 hours after the intervention
  The time of first use of rescue analgesia
First time out-of-bed | From date of surgery until the date of first out-of-bed，assessed up to 7 days
  Time of participant's first out-of-bed activity after surgery
Length of hospital stay | From date of surgery until the date of first hospital discharge，assessed up to 1 months
  Duration of participants from hospital admission to hospital discharge
Chronic pain score | postoperative day (POD) 90
  Use pain Numeric Rating Scale(NRS) to evaluate the movement-evoked pain score and rest pain score at 90 days after surgery.(NRS scale 0-10, where 0 was no pain, and 10 was the worst possible pain)
Score of satisfaction with analgesia | At 72 hours after the intervention
  At 72 hours after the intervention,the participants rated the satisfaction with analgesia.Satisfaction rating scale 0-5,where 0 was poor drug effectiveness, and 5 was excellent drug efficacy)

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, ph.D, Study Chair — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China